CLINICAL TRIAL: NCT05755230
Title: My Journey - Prospective Cohort of Perioperative Results
Brief Title: Prospective Cohort of Perioperative Results
Status: Recruiting | Type: Observational
Sponsor: COPAL - My Journey (Network)
Responsible Party: Principal Investigator, Santiago Mc Loughlin, MD, COPAL - My Journey
Other Study IDs: 1-Copal
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Perioperative/Postoperative Complications
Keywords: Periopererative; Enhanced Recovery
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Perioperative online register of the care process and outcomes. Observational prospective cohort.

DETAILED DESCRIPTION:
Center are invited to join the perioperative register where they input anonymized data about the surgical process and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2043-01-01 (Estimated); Study Completion 2050-01-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative International Register | 20 years
  Collaborative register of preoperative variables

CONTACTS AND LOCATIONS:
Locations (1):
- COPAL, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided